CLINICAL TRIAL: NCT03956667
Title: Music:ED iMpact of therapeUtic Live muSic on Pain and Distress Levels During Interventions Within the paediatriC Emergency Department
Brief Title: iMpact of therapeUtic Live muSic on Pain and Distress Levels During Interventions in the paediatriC Emergency Department
Acronym: Music:ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 225890
Record Dates: First submitted 2019-01-09; First posted 2019-05-21 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: Paediatric; distress; Paediatric Emergency Department; Music
MeSH Terms: conditions — Pain

STUDY DESIGN:
Masking Description: Participants will be recruited to the experimental (Live Music) arm on days that the musicians are working in the Emergency Department.
  Participants will be recruited to the control (Non Music) arm on days that there are no musicians present in the Emergency Department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Live Music (Experimental): Live Music will be played during the required Emergency Department procedure.
  Interventions: Other: Live Music
- Control: No Live Music (No Intervention): There will be no music played during the required Emergency Department procedure.

INTERVENTIONS:
Other: Live Music — Musicians from Cascade Music will provide recruited participants in the experimental arm with high-quality calming, distracting music during their Emergency Department procedure.
  Arms: Experimental: Live Music

SUMMARY:
The Emergency Department (ED) can be stressful and traumatic, especially for children and young people, and the clinical environment can be a frightening, unfamiliar space, which adds to an already anxious experience.

Musicians from Cascade Music, who have an established track record of working with the Paediatric ED, will provide recruited participants in the experimental arm with high-quality calming, distracting music during selected procedures. A wide range of music will be used, ranging from nursery rhymes to classical to pop tunes, to engage with and comfort children, taking their attention away from their immediate pain or distress. Pain scores throughout the procedure will be self-assessed by patients (if old enough to use a self assessment tool i.e. 3 years and above) as well as observed by a Research Nurse. Qualitative data on distress and the experiences of patients, families and staff will also be collected via a questionnaire. Participants recruited to the control arm will complete the same measures but receive no live music.

This project is underpinned by three areas of need:

1. Despite there being a wide breadth of clinical studies that have used music within various healthcare settings, one area that has been almost completely unexplored is the Paediatric Emergency Department (PED). Alder Hey Children's Hospital (AHCH), as a world leader in research, is ideally situated to conduct this preliminary research.
2. By 2020 AHCH plans to be a world class, child-focused centre of research, innovation and education expertise to improve the health and wellbeing outcomes for children and young people. Supporting patients through stressful and invasive procedures is crucial. Inspired by the patients and families that we care for, this research fits well with the AHCH vision, demonstrating an innovative and evidence-informed approach to enhancing practice.
3. The University of Liverpool's impact intensive approach to research is a key strength. This study is designed to have a positive immediate impact on the children and young people participating and those undergoing interventional procedures in the future, helping to enhance patient experience of the ED.

DETAILED DESCRIPTION:
Value of the study:

There is a growing evidence-base for the use of music in healthcare settings, with music already demonstrated to reduce stress, distress and the perception of pain in some clinical contexts. Yet, there is a lack of studies examining the impact of live music in paediatric emergency contexts.

A literature review revealed that there is a lack of studies examining the impact of live music in paediatric emergency contexts.

Related studies either used recorded music in the place of live music, or, if live music was used, then it was within a non-emergency setting.

The Music:ED study will therefore use a controlled experimental design to investigate the impact of using therapeutic live music in the Alder Hey Paediatric Emergency Department to reduce pain and distress during interventional procedures.

The outcomes of the study will provide evidence for the use of live music in the PED to support and enhance patient experience. Distress is often particularly high within the emergency department. If a patient's experience whilst attending the Emergency Department can be less traumatic, this will be of benefit to all: patients, families and clinicians. A patient who is less distressed is more cooperative and may be easier and quicker to treat.

Methodology and Methods

Research Question:

Does live music decrease the pain and distress of patients undergoing a procedure within the paediatric emergency department?

Aims of the Study:

The aims/objectives include:

1. To explore whether live music helps to decrease pain and distress in patients in the Paediatric Emergency Department
2. To explore whether procedures can be carried out with greater ease from a clinician's perspective and whether staff experience of the situation is impacted by the presence of live music.
3. Exploring the overall impact on the ED experience from the patients, families and clinicians' perspectives.

Methodological Approach:

A mixed method design has been chosen to provide the investigators with different forms of data and insights from multiple practitioner, parent and patient perspectives throughout the experience.

Quantitative data includes collecting information about the patient's pain levels using both self-assessed pain scores (Wong Baker scoring) and assessed pain scores (FLACC pain tool).

Qualitative data will be collected from open response questionnaires to explore patient distress and the practitioner, parent and patient perspectives on the experience.

Methods:

There will be an experimental (live music) and a control (no live music) group. Research Nurses will identify appropriate patients using a screening tool that will outline the inclusion/exclusion criteria. Participant Information Sheets (PIS) will be provided to patients and their families for their appropriate ages. They will be offered a copy of the results if they would like and will be told how the results will be reported when the study is completed.

After gaining written consent from the parent and written or verbal assent from the child, Wong-Baker pain scoring methods will be explained in advance of the procedure.

Necessary data will be collected for the Case Report Form (CRF).

The participant's involvement in the study will be limited to the length of time of their Emergency Department visit, so will be just one day and one procedure.

For the experimental (music) group, Cascade's musicians will spend eight weeks, twelve hours per week in the ED and will aim to recruit all eligible children during that period. As this is a pilot study recruitment targets need to remain flexible, but are estimated at 60-80 participants (per group).

The same number of participants will be recruited to the control (no live music) group as a comparison, on days that the musicians are not in the department. All patients in both groups will continue to receive standard care. Each child can only be in the study once and for one procedure. Patients will be free to withdraw from the study at any time.

Following the procedure and interviews, patients involved will be offered a sticker and a CD of calming music recorded by Cascade Music as a thank you for their participation. For ethical reasons, this will not be mentioned in advance.

Methods of data collection and analysis

Three sets of data will be collected:

1. Quantitative: Self-reported pain. A validated observational tool will be used: Wong Baker Faces. This is suitable for children age 3+. As children self-report, the Research Nurse will collect this data on a paper CRF. Wong Baker scores will be collected before, during and after the procedure. If mid-procedure collection of pain score is inappropriate, then participants can be asked about mid-procedure pain scores after the procedure.

   A self-reported pain score will also be taken in advance, during the recruitment process, to provide a baseline measure.
2. Quantitative: Observed pain. Data will be collected on observed pain levels using a validated observational tool: Faces, Legs, Activity, Cry and Consolability (FLACC) pain assessment tool.

   This tool is suitable and validated for all ages of the recruited participants, from 6 months until 16 years. References regarding justification of this scale for these age ranges are below.

   Scoring will take place before, during and after the procedure. The Research Nurse will carry out this scoring, and when available, an independent observer from the Emergency Department staff will also. The Research Nurse will collect this data on the paper CRF.

   Heart rate will also be monitored throughout, where a child is cooperative enough. HR will be noted approximately every two minutes before, during and after procedure, (cleaning marks the beginning of the procedure, final bandage/dressing marks the completion). The Research Nurse will note HR data on the CRF. There will be an option for the Research Nurse to record 'not available' for heart rate measurements either because child refuses or because of probe or monitor issues etc.
3. Qualitative: Distress and experiences of patients, families and clinicians. Outcome measures will include collecting qualitative information on patient's distress, and patients', families' and clinician's Emergency Department experience. All recruited patients will receive a paper questionnaire with open text response options.

Qualitative questions for Experimental AND Control Groups:

The following two questions will be asked of both the experimental (live music) AND control (no live music) groups. The questions will be asked of each of these two people: patient and parent/legal guardian.

'Please answer the following questions, in particular, in regard to distress levels/lack of distress':

* Qualitative question 1. What do you think helped you/your child during their procedure?
* Qualitative question 2. Did anything make the situation worse?

Qualitative questions for Experimental Group Only:

Within the experimental group only, the following three additional questions will be asked, via a paper questionnaire, of each of these three people: patient, parent/legal guardian and clinician. These questions directly link to the objectives of the study.

These questions are in particular regard to music, which is why they would not be appropriate to be asked of the control (no live music) group.

* Qualitative Question 1. How did you feel the music affected the child's distress before, during and after the procedure?
* Qualitative Question 2. Can you tell me about how the live music helped or hindered the procedure?
* Qualitative Question 3. Can you tell me about your experience of the ED (Emergency Department) today, in particular in regard to the music?

The qualitative questions will be included in a open ended questionnaire style sheet which the parent, child or practitioner if the parent wishes, can fill out between the end of the music intervention and when they are discharged from the ward. It will be collected by the RN and stored in a secure room in a locked filing cabinet.

Target population and sampling This will be a single centre study. Study participants for both the control and experimental groups of the study will be recruited from AHCH Emergency Department. The study population will consist of children between the age of 6 months and 16 years needing to undergo a painful procedure from a specified list. The Research Nurse will use a screening tool to assess eligibility within this age group.

Necessary data will be collected for the CRF (Case Report Form) by the Research Nurse:

CRF:

* Patient's name
* Patient's age
* Patient's gender
* Parent(s)/legal guardian in attendance during procedure (names)
* Whether or not the patient has had this procedure before
* How many times the child has visited the hospital in the last 12 months
* Have they had an upsetting hospital experience in the past? Yes or no
* Record a Wong-Baker pain score at this point (for children age 3+) as a baseline measure
* Record whether patient has had analgesia in advance, or during hospital visit
* Record use of local anaesthetics e.g EMLA/ametop, LAT gel, cold spray (ethyl chloride)
* Record use of Entonox during the procedure
* Record if other distraction methods were also used (Play Specialist/books/bubbles/IPad/TV/ IPhone/ staff dancing and singing, etc)
* Record whether the procedure was successful
* Record the duration of the procedure (cleaning marks the beginning of the procedure, final bandage/dressing marks the completion)
* Record how many attempts were required to carry out procedure
* Record the role and grade of the Clinician carrying out the procedure
* Record heart rate at 2-minute intervals if tolerated. Include option for the research nurse to record 'not available' for heart rate measurements either because child refuses or if probe or monitor issues etc
* Record whether there is an independent observer present. If so, who?

ELIGIBILITY:
Inclusion Criteria:

* Parent/Legal Guardian present and able to consent.
* Age range: 6 months - 16 years.
* Procedures: Capillary blood sampling, cannulation, venepuncture, suturing, wound cleaning and closure.
* Families and children whose primary language is other than English will be included in the study if their English speaking skills are at a level that they can understand and complete the consent/assent process.

Exclusion Criteria:

* Children with Special Educational Needs, children with global development delay, sensory impairments, neurological deficits or disorders, impairment to pain i.e. spina bifida.
* Children in resuscitation or unconscious.
* Non-English speaking.
* Suspected ingestion of recreational drugs, antidepressants or alcohol
* Concerns relating to NAI (non accidental injury)/safeguarding concerns
* Life or limb critical injuries
* Children too unwell to participate

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Lower Self-Reported Pain scores in the Interventional Arm. | One day
  Participants' Self-Reported pain scores will be noted by the Research Nurse using the Wong-Baker pain scoring tool. Scores will be collected before, during and after the procedure.
Lower Observed Pain scores in the Interventional Arm. | One day
  Observed Pain scores will be observed and collected by the Research Nurse using the FLACC (Faces, Legs, Activity, Cry and Consolability) pain scoring tool.
  FLACC Scoring will take place before, during and after the procedure.

SECONDARY OUTCOMES:
Lower distress levels recorded in qualitative data collection in the interventional arm. | One day
  Qualitative questions will be asked via a paper questionnaire regarding distress levels and experiences of patients, families and clinicians
Reduced heart rates in the interventional compared to the control arm. | One day
  Heart rate will be monitored throughout as an additional marker, where a child is cooperative enough. HR will be noted approximately every two minutes before, during and after procedure, (cleaning marks the beginning of the procedure, final bandage/dressing marks the completion). The Research Nurse will note HR data on the CRF. There will be an option for the Research Nurse to record 'not available' for heart rate measurements either because child refuses or because of probe or monitor issues etc.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Durand, MBChBMRCPCH, Principal Investigator — Alder Hey Children's NHS Foundation Trust
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT03956667/Prot_000.pdf